CLINICAL TRIAL: NCT04251247
Title: Diagnostic Value of D-dimer/Fibrinogen Ratio in Patients With Acute Aortic Dissection
Status: Recruiting | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Can Topcu, Director of Department of Cardiovascular Surgery, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2020/514/169/B
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Aortic Dissection; Pulmonary Embolism
MeSH Terms: conditions — Aortic Dissection; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute aortic dissection: Patients with a diagnosis of acute aortic dissection.
  Interventions: Diagnostic Test: D-dimer/fibrinogen ratio
- Acute pulmonary embolism: Patients with a diagnosis of acute pulmonary embolism
  Interventions: Diagnostic Test: D-dimer/fibrinogen ratio
- Non-cardiac chest pain: Patients with non-cardiac chest pain
  Interventions: Diagnostic Test: D-dimer/fibrinogen ratio

INTERVENTIONS:
Diagnostic Test: D-dimer/fibrinogen ratio — The ratio of D-dimer (ng/ml) to fibrinogen (mg/dl)

SUMMARY:
Acute aortic dissection is rare but potentially life-threatening disease with an incidence of 5-30 cases per million, annually. Therefore prompt diagnosis is crucial. D-dimer values have been shown to be useful in the diagnosis of acute aortic dissection. Fibrinogen levels have been shown to be low, normal or high in individuals with acute aortic dissection. This study aims to investigate whether D-dimer/fibrinogen ratio can be valuable for diagnosis of acute aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute aortic dissection
* Diagnosis of acute pulmonary embolism
* Diagnosis of non-cardiac chest pain

Exclusion Criteria:

* Any etiology of chest pain other than acute aortic dissection, acute pulmonary embolism, or non-cardiac chest pain
* Participants who do not give consent for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to emergency department with chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Acute aortic dissection | 24 hours
  Diagnosis of acute aortic dissection confirmed by contrast enhanced computed tomography, magnetic resonance imaging, echocardiography or aortography

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul
  - Kartal Dr. Lutfi Kirdar Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hajsadeghi S, Kerman SR, Khojandi M, Vaferi H, Ramezani R, Jourshari NM, Mousavi SA, Pouraliakbar H. Accuracy of D-dimer:fibrinogen ratio to diagnose pulmonary thromboembolism in patients admitted to intensive care units. Cardiovasc J Afr. 2012 Sep;23(8):446-56. doi: 10.5830/CVJA-2012-041. PMID 23044500
- [Background] Kara H, Bayir A, Degirmenci S, Kayis SA, Akinci M, Ak A, Celik B, Dogru A, Ozturk B. D-dimer and D-dimer/fibrinogen ratio in predicting pulmonary embolism in patients evaluated in a hospital emergency department. Acta Clin Belg. 2014 Aug;69(4):240-5. doi: 10.1179/2295333714Y.0000000029. PMID 25012747
- [Background] Guan XL, Wang XL, Liu YY, Lan F, Gong M, Li HY, Liu O, Jiang WJ, Liu YM, Zhu JM, Sun LZ, Zhang HJ. Changes in the Hemostatic System of Patients With Acute Aortic Dissection Undergoing Aortic Arch Surgery. Ann Thorac Surg. 2016 Mar;101(3):945-51. doi: 10.1016/j.athoracsur.2015.08.047. Epub 2015 Oct 23. PMID 26603023
- [Background] Eggebrecht H, Naber CK, Bruch C, Kroger K, von Birgelen C, Schmermund A, Wichert M, Bartel T, Mann K, Erbel R. Value of plasma fibrin D-dimers for detection of acute aortic dissection. J Am Coll Cardiol. 2004 Aug 18;44(4):804-9. doi: 10.1016/j.jacc.2004.04.053. PMID 15312863